CLINICAL TRIAL: NCT03902899
Title: The Influence of a Short Training in the Detection Rate of Proximal Serrated Polyps in an Asymptomatic Patient Population
Brief Title: Increasing Serrated Polyp Detection With a Brief Awareness Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DW18001
Record Dates: First submitted 2019-01-04; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Serrated Polyp; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a non-randomized controlled trial with two arms. The intervention-arm consists of all endoscopists employed by 9 semi-randomly chosen Dutch hospitals hospitals who receive an educational training. The control-arm consists of a specific number of randomly chosen endoscopists.
Masking Description: The investigator personally delivers the training and can thus not be blinded for the endoscopists allocated to the intervention-arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-arm (Experimental): All endoscopists employed by 9 semi-randomly chosen hospitals in the Netherlands will be exposed to an educational intervention (oral presentation): an oral awareness training which will be delivered twice, first in 2014 and then in 2016/2017.
  In total 38 endoscopists are included from these 9 hospitals.
  Interventions: Other: Educational intervention (oral presentation)
- Control arm (No Intervention): A random set of 100 endoscopists will be selected ass a reference group. These 100 endoscopists were unaware of the present study, and were thus blinded for their allocation.

INTERVENTIONS:
Other: Educational intervention (oral presentation) — A brief oral presentation (30-45 minutes) which focused on making endoscopists aware of the significance and characteristics of serrated polyps.
  Arms: Intervention-arm

SUMMARY:
In this non-randomized controlled trial, a semi-random group of Dutch endoscopist receive an oral training about the significance of serrated polyps. The primary aim of this training is to improve the endoscopist's awareness of the significance of serrated polyps, ultimately leading to increased detection. In addition, a random group of endoscopists that will not receive this training will be used as a reference group.

Data will be collected as part of routine care within the Nationwide Dutch Bowel cancer screening program. The serrated polyp detectionrate of each endoscopist will be extracted from anonymized data that will be prospectively collected as part of routine care within the Dutch Nationwide bowel cancer screening program. Data will be anonymized and provided by Rijksinstituut voor Volksgezondheid en Milieu (RIVM) and ScreenIT.

ELIGIBILITY:
Inclusion criteria:

- Endoscopists accredited to perform colonoscopies within the Dutch Nationwide colorectal cancer screening program

Exclusion criteria:

- Absent during both training sessions while employed in one of the trained hospitals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Proximal serrated polyp detection rate (PSPDR) | Up to five years (between 2014 and 2018)
  Rate/proportion of an endoscopist's colonoscopies with one or more serrated polyps proximal to or in splenic flexure.

SECONDARY OUTCOMES:
Adenoma detection rate (ADR) | Up to five years (between 2014 and 2018)
  Rate/proportion of an endoscopist's colonoscopies with one or more adenomas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bleijenberg AGC, van Leerdam ME, Bargeman M, Koornstra JJ, van Herwaarden YJ, Spaander MC, Sanduleanu S, Bastiaansen BAJ, Schoon EJ, van Lelyveld N, Dekker E, IJspeert JEG. Substantial and sustained improvement of serrated polyp detection after a simple educational intervention: results from a prospective controlled trial. Gut. 2020 Dec;69(12):2150-2158. doi: 10.1136/gutjnl-2019-319804. Epub 2020 Mar 5. PMID 32139550